CLINICAL TRIAL: NCT04761744
Title: A Phase II Study of Nivolumab in Patients With Genetic Alterations in DNA Damage Repair and Response Who Progressed After Standard Treatment for Metastatic Solid Cancers
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korean Cancer Study Group (Other)
Responsible Party: Principal Investigator, Kyong-Hwa, Park, Professor, Korean Cancer Study Group
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KM-06
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: DDR Gene Mutation; Metastatic Solid Tumor
Keywords: Nivolumab
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nivolumab (Experimental)
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Study treatment consists of nivolumab 3mg/kg, and will be repeated every 2 weeks.

SUMMARY:
A Phase II Study of Nivolumab in Patients with Genetic alterations in DNA Damage repair and response Who Progressed after Standard treatment for Metastatic Solid Cancers

DETAILED DESCRIPTION:
All the patients will be included in the final analysis, with a total of 48 patients to be enrolled.

Treatment will occur until disease progression, unacceptable toxicity or patient withdrawal.

Study treatment consists of nivolumab 3mg/kg, and will be repeated every 2 weeks.

Response evaluation will be performed every 6 weeks (+/- 1 week window period is allowed).

ELIGIBILITY:
Inclusion Criteria:

1. Patient has histologically and/or cytologically confirmed diagnosis of cancers in colon, stomach, biliary tract, breast, bladder and upper urinary tract, endometrium, ovarian, prostate, and other cancers.
2. Alterations in DNA damage repair and response genes assessed by next-generation sequencing (K-MASTER panel assay of ≥370 genes)
3. Progressed after at least first-line systemic chemotherapy for metastatic setting.
4. ≥ 1 measurable lesion(s) by RECIST 1.1.
5. Unresectable advanced or metastatic disease.
6. Age over 20 years old.
7. ECOG 0-1, but final decision by clinical.
8. Adequate organ functions.

   1. Bone marrow function: Hemoglobin ≥ 9.0 g/dL, ANC ≥ 1,500/mm3, platelet ≥ 100,000/mm3
   2. Hepatic functions: bilirubin ≤ 1.5 X ULN, AST/ALT ≤ 2.5 X ULN (≤ 5 X ULN in cases of liver metastasis)
   3. Renal functions: serum Cr ≤ 1.5 X ULN or calculated CCr (Cockroft) ≥ 30 ml/min
9. Be willing and able to comply with the protocol for the duration of the study.
10. Give written informed consent prior to study-specific screening procedures, with the understanding that the patient has the right to withdraw the study at any time, without prejudice.
11. Female subjects must either be of non-reproductive potential (≥ 60 years old and no menses for ≥ 1 year without an alternative medical cause, or history of hysterectomy, or history of bilateral tubal ligation, or history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry.
12. Women of childbearing potential and men must agree to use highly efficient contraception since signing of the IC form until at least 6 Month after the last study drug administration.

Exclusion Criteria:

1. Any prior treatment with PD-1 or PD-L1 inhibitor.
2. Receipt of the last dose of chemotherapy ≤ 28 days prior to the first dose of study drugs.
3. Current or prior use of immunosuppressive medication within 28 days before the first dose of nivolumab, with the exceptions for the following:

   1. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection);
   2. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent;
   3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
4. Concurrent or previous history of another primary cancer within 3 years prior to randomization except for curatively treated cervical cancer in situ, non-melanomatous skin cancer, superficial bladder cancer (pTis and pT1) and curatively treated thyroid cancer of any stage. Concurrent, histologically confirmed, unresected thyroid cancer without distant metastasis could be allowed with the agreement of the chief principal investigator.
5. Uncontrolled CNS metastases; permitted if asymptomatic or neurologically stable.
6. Prior radiation therapy would be permitted, but non-radiated evaluable lesions should be present at study entry.
7. Radiation therapy during study treatment is not permitted, but if the local investigator decides that radiation therapy should be given during study treatments, he should be convinced that there is no evidence of disease progression with agreement of the chief principal investigator.
8. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
9. Active or prior documented autoimmune disease within the past 2 years; subjects with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible.
10. Active or prior documented inflammatory bowel disease.
11. History of prior immunodeficiency.
12. History of allogeneic organ transplantation.
13. Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v4.03 Grade ≥ 3)
14. Clinical diagnosis of active tuberculosis.
15. Vaccination within 4 weeks of the first dose of nivolumab and while on trials is prohibited except for administration of inactivated vaccines
16. Known history of testing positive for HIV
17. Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive). Except, resolved HBV infection (as evidenced by detectable HBV surface antibody, detectable HBV core antibody, undetectable HBV DNA, and undetectable HBV surface antigen) or Chronic HBV infection (as evidenced by detectable HBV surface antigen or HBV DNA). Subjects with chronic HBV infection must have HBV DNA <100IU/ml and must be on antiviral therapy)
18. Major surgery or significant traumatic injury within 28 days prior to study treatment.
19. Non-healing wound, ulcer, or bone fracture.
20. Current evidence of significant gastrointestinal bleeding or (impending) obstruction.
21. Concomitant participation in another clinical trial.
22. Pregnant of breast-feeding subjects. Women of child-bearing potential must have pregnancy test within 7 days and a negative result must be documented before start of study treatment.
23. Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results.
24. Active infection requiring systemic therapy.
25. Persisting toxicity related to prior therapy (NCI CTCAE v. 4.03 Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable.
26. Other severe acute or chronic medical conditions including colitis, inflammatory bowel disease, pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
27. Patient who can't comply with the protocol and who is not willing to comply with the protocol.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-06-14 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | within maximum 3 years
  the percentage of patients experiencing confirmed complete response (CR) and partial response (PR) assessed by RECIST criteria v.1.1

SECONDARY OUTCOMES:
Progression free survival | within maximum 3 years
  the time from study entry until the first observation of disease progression
Overall survival | within maximum 3 years
  the time from study entry until death

CONTACTS AND LOCATIONS:
Overall Officials: Kyong Hwa Park, MD, PhD, Principal Investigator — Korean Cancer Study Group
Locations (2):
- South Korea (2):
  - Korean Cancer Study Group, Seoul, Chongro-ku
  - Korea University Anam Hospital, Seoul, Seongbuk-gu, Inchon-ro

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oldham RK. Biologicals and biological response modifiers: fourth modality of cancer treatment. Cancer Treat Rep. 1984 Jan;68(1):221-32. PMID 6198081
- [Background] Waldmann TA. Immunotherapy: past, present and future. Nat Med. 2003 Mar;9(3):269-77. doi: 10.1038/nm0303-269. No abstract available. PMID 12612576
- [Background] Borghaei H, Paz-Ares L, Horn L, Spigel DR, Steins M, Ready NE, Chow LQ, Vokes EE, Felip E, Holgado E, Barlesi F, Kohlhaufl M, Arrieta O, Burgio MA, Fayette J, Lena H, Poddubskaya E, Gerber DE, Gettinger SN, Rudin CM, Rizvi N, Crino L, Blumenschein GR Jr, Antonia SJ, Dorange C, Harbison CT, Graf Finckenstein F, Brahmer JR. Nivolumab versus Docetaxel in Advanced Nonsquamous Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Oct 22;373(17):1627-39. doi: 10.1056/NEJMoa1507643. Epub 2015 Sep 27. PMID 26412456
- [Background] Ferris RL, Blumenschein G Jr, Fayette J, Guigay J, Colevas AD, Licitra L, Harrington K, Kasper S, Vokes EE, Even C, Worden F, Saba NF, Iglesias Docampo LC, Haddad R, Rordorf T, Kiyota N, Tahara M, Monga M, Lynch M, Geese WJ, Kopit J, Shaw JW, Gillison ML. Nivolumab for Recurrent Squamous-Cell Carcinoma of the Head and Neck. N Engl J Med. 2016 Nov 10;375(19):1856-1867. doi: 10.1056/NEJMoa1602252. Epub 2016 Oct 8. PMID 27718784
- [Background] Larkin J, Chiarion-Sileni V, Gonzalez R, Grob JJ, Cowey CL, Lao CD, Schadendorf D, Dummer R, Smylie M, Rutkowski P, Ferrucci PF, Hill A, Wagstaff J, Carlino MS, Haanen JB, Maio M, Marquez-Rodas I, McArthur GA, Ascierto PA, Long GV, Callahan MK, Postow MA, Grossmann K, Sznol M, Dreno B, Bastholt L, Yang A, Rollin LM, Horak C, Hodi FS, Wolchok JD. Combined Nivolumab and Ipilimumab or Monotherapy in Untreated Melanoma. N Engl J Med. 2015 Jul 2;373(1):23-34. doi: 10.1056/NEJMoa1504030. Epub 2015 May 31. PMID 26027431
- [Background] Motzer RJ, Escudier B, McDermott DF, George S, Hammers HJ, Srinivas S, Tykodi SS, Sosman JA, Procopio G, Plimack ER, Castellano D, Choueiri TK, Gurney H, Donskov F, Bono P, Wagstaff J, Gauler TC, Ueda T, Tomita Y, Schutz FA, Kollmannsberger C, Larkin J, Ravaud A, Simon JS, Xu LA, Waxman IM, Sharma P; CheckMate 025 Investigators. Nivolumab versus Everolimus in Advanced Renal-Cell Carcinoma. N Engl J Med. 2015 Nov 5;373(19):1803-13. doi: 10.1056/NEJMoa1510665. Epub 2015 Sep 25. PMID 26406148
- [Background] Francisco LM, Sage PT, Sharpe AH. The PD-1 pathway in tolerance and autoimmunity. Immunol Rev. 2010 Jul;236:219-42. doi: 10.1111/j.1600-065X.2010.00923.x. PMID 20636820
- [Background] Okazaki T, Honjo T. The PD-1-PD-L pathway in immunological tolerance. Trends Immunol. 2006 Apr;27(4):195-201. doi: 10.1016/j.it.2006.02.001. Epub 2006 Feb 24. PMID 16500147
- [Background] Zou W, Chen L. Inhibitory B7-family molecules in the tumour microenvironment. Nat Rev Immunol. 2008 Jun;8(6):467-77. doi: 10.1038/nri2326. PMID 18500231
- [Background] Hamanishi J, Mandai M, Iwasaki M, Okazaki T, Tanaka Y, Yamaguchi K, Higuchi T, Yagi H, Takakura K, Minato N, Honjo T, Fujii S. Programmed cell death 1 ligand 1 and tumor-infiltrating CD8+ T lymphocytes are prognostic factors of human ovarian cancer. Proc Natl Acad Sci U S A. 2007 Feb 27;104(9):3360-5. doi: 10.1073/pnas.0611533104. Epub 2007 Feb 21. PMID 17360651
- [Background] Hino R, Kabashima K, Kato Y, Yagi H, Nakamura M, Honjo T, Okazaki T, Tokura Y. Tumor cell expression of programmed cell death-1 ligand 1 is a prognostic factor for malignant melanoma. Cancer. 2010 Apr 1;116(7):1757-66. doi: 10.1002/cncr.24899. PMID 20143437
- [Background] Ohigashi Y, Sho M, Yamada Y, Tsurui Y, Hamada K, Ikeda N, Mizuno T, Yoriki R, Kashizuka H, Yane K, Tsushima F, Otsuki N, Yagita H, Azuma M, Nakajima Y. Clinical significance of programmed death-1 ligand-1 and programmed death-1 ligand-2 expression in human esophageal cancer. Clin Cancer Res. 2005 Apr 15;11(8):2947-53. doi: 10.1158/1078-0432.CCR-04-1469. PMID 15837746
- [Background] Thompson RH, Kuntz SM, Leibovich BC, Dong H, Lohse CM, Webster WS, Sengupta S, Frank I, Parker AS, Zincke H, Blute ML, Sebo TJ, Cheville JC, Kwon ED. Tumor B7-H1 is associated with poor prognosis in renal cell carcinoma patients with long-term follow-up. Cancer Res. 2006 Apr 1;66(7):3381-5. doi: 10.1158/0008-5472.CAN-05-4303. PMID 16585157
- [Background] Nomi T, Sho M, Akahori T, Hamada K, Kubo A, Kanehiro H, Nakamura S, Enomoto K, Yagita H, Azuma M, Nakajima Y. Clinical significance and therapeutic potential of the programmed death-1 ligand/programmed death-1 pathway in human pancreatic cancer. Clin Cancer Res. 2007 Apr 1;13(7):2151-7. doi: 10.1158/1078-0432.CCR-06-2746. PMID 17404099
- [Background] Nakanishi J, Wada Y, Matsumoto K, Azuma M, Kikuchi K, Ueda S. Overexpression of B7-H1 (PD-L1) significantly associates with tumor grade and postoperative prognosis in human urothelial cancers. Cancer Immunol Immunother. 2007 Aug;56(8):1173-82. doi: 10.1007/s00262-006-0266-z. Epub 2006 Dec 22. PMID 17186290
- [Background] Rizvi NA, Hellmann MD, Snyder A, Kvistborg P, Makarov V, Havel JJ, Lee W, Yuan J, Wong P, Ho TS, Miller ML, Rekhtman N, Moreira AL, Ibrahim F, Bruggeman C, Gasmi B, Zappasodi R, Maeda Y, Sander C, Garon EB, Merghoub T, Wolchok JD, Schumacher TN, Chan TA. Cancer immunology. Mutational landscape determines sensitivity to PD-1 blockade in non-small cell lung cancer. Science. 2015 Apr 3;348(6230):124-8. doi: 10.1126/science.aaa1348. Epub 2015 Mar 12. PMID 25765070
- [Background] Balar AV, Galsky MD, Rosenberg JE, Powles T, Petrylak DP, Bellmunt J, Loriot Y, Necchi A, Hoffman-Censits J, Perez-Gracia JL, Dawson NA, van der Heijden MS, Dreicer R, Srinivas S, Retz MM, Joseph RW, Drakaki A, Vaishampayan UN, Sridhar SS, Quinn DI, Duran I, Shaffer DR, Eigl BJ, Grivas PD, Yu EY, Li S, Kadel EE 3rd, Boyd Z, Bourgon R, Hegde PS, Mariathasan S, Thastrom A, Abidoye OO, Fine GD, Bajorin DF; IMvigor210 Study Group. Atezolizumab as first-line treatment in cisplatin-ineligible patients with locally advanced and metastatic urothelial carcinoma: a single-arm, multicentre, phase 2 trial. Lancet. 2017 Jan 7;389(10064):67-76. doi: 10.1016/S0140-6736(16)32455-2. Epub 2016 Dec 8. PMID 27939400
- [Background] Teo MY, Seier K, Ostrovnaya I, Regazzi AM, Kania BE, Moran MM, Cipolla CK, Bluth MJ, Chaim J, Al-Ahmadie H, Snyder A, Carlo MI, Solit DB, Berger MF, Funt S, Wolchok JD, Iyer G, Bajorin DF, Callahan MK, Rosenberg JE. Alterations in DNA Damage Response and Repair Genes as Potential Marker of Clinical Benefit From PD-1/PD-L1 Blockade in Advanced Urothelial Cancers. J Clin Oncol. 2018 Jun 10;36(17):1685-1694. doi: 10.1200/JCO.2017.75.7740. Epub 2018 Feb 28. PMID 29489427
- [Background] Mouw KW, Goldberg MS, Konstantinopoulos PA, D'Andrea AD. DNA Damage and Repair Biomarkers of Immunotherapy Response. Cancer Discov. 2017 Jul;7(7):675-693. doi: 10.1158/2159-8290.CD-17-0226. Epub 2017 Jun 19. PMID 28630051
- [Background] Lawrence MS, Stojanov P, Mermel CH, Robinson JT, Garraway LA, Golub TR, Meyerson M, Gabriel SB, Lander ES, Getz G. Discovery and saturation analysis of cancer genes across 21 tumour types. Nature. 2014 Jan 23;505(7484):495-501. doi: 10.1038/nature12912. Epub 2014 Jan 5. PMID 24390350
- [Background] Jung HA, Park YH, Kim M, Kim S, Chang WJ, Choi MK, Hong JY, Kim SW, Kil WH, Lee JE, Nam SJ, Ahn JS, Im YH. Prognostic relevance of biological subtype overrides that of TNM staging in breast cancer: discordance between stage and biology. Tumour Biol. 2015 Feb;36(2):1073-9. doi: 10.1007/s13277-014-2730-2. Epub 2014 Oct 19. PMID 25326808
- [Background] Burrell RA, McGranahan N, Bartek J, Swanton C. The causes and consequences of genetic heterogeneity in cancer evolution. Nature. 2013 Sep 19;501(7467):338-45. doi: 10.1038/nature12625. PMID 24048066
- [Background] Kelderman S, Schumacher TN, Kvistborg P. Mismatch Repair-Deficient Cancers Are Targets for Anti-PD-1 Therapy. Cancer Cell. 2015 Jul 13;28(1):11-3. doi: 10.1016/j.ccell.2015.06.012. PMID 26175412
- [Background] Le DT, Uram JN, Wang H, Bartlett BR, Kemberling H, Eyring AD, Skora AD, Luber BS, Azad NS, Laheru D, Biedrzycki B, Donehower RC, Zaheer A, Fisher GA, Crocenzi TS, Lee JJ, Duffy SM, Goldberg RM, de la Chapelle A, Koshiji M, Bhaijee F, Huebner T, Hruban RH, Wood LD, Cuka N, Pardoll DM, Papadopoulos N, Kinzler KW, Zhou S, Cornish TC, Taube JM, Anders RA, Eshleman JR, Vogelstein B, Diaz LA Jr. PD-1 Blockade in Tumors with Mismatch-Repair Deficiency. N Engl J Med. 2015 Jun 25;372(26):2509-20. doi: 10.1056/NEJMoa1500596. Epub 2015 May 30. PMID 26028255
- [Background] Parikh AR, He Y, Hong TS, Corcoran RB, Clark JW, Ryan DP, Zou L, Ting DT, Catenacci DV, Chao J, Fakih M, Klempner SJ, Ross JS, Frampton GM, Miller VA, Ali SM, Schrock AB. Analysis of DNA Damage Response Gene Alterations and Tumor Mutational Burden Across 17,486 Tubular Gastrointestinal Carcinomas: Implications for Therapy. Oncologist. 2019 Oct;24(10):1340-1347. doi: 10.1634/theoncologist.2019-0034. Epub 2019 Apr 30. PMID 31040255
- [Background] Strickland KC, Howitt BE, Shukla SA, Rodig S, Ritterhouse LL, Liu JF, Garber JE, Chowdhury D, Wu CJ, D'Andrea AD, Matulonis UA, Konstantinopoulos PA. Association and prognostic significance of BRCA1/2-mutation status with neoantigen load, number of tumor-infiltrating lymphocytes and expression of PD-1/PD-L1 in high grade serous ovarian cancer. Oncotarget. 2016 Mar 22;7(12):13587-98. doi: 10.18632/oncotarget.7277. PMID 26871470
- [Background] Colebatch A, Hitchins M, Williams R, Meagher A, Hawkins NJ, Ward RL. The role of MYH and microsatellite instability in the development of sporadic colorectal cancer. Br J Cancer. 2006 Nov 6;95(9):1239-43. doi: 10.1038/sj.bjc.6603421. Epub 2006 Oct 10. PMID 17031395
- [Background] Hugo W, Zaretsky JM, Sun L, Song C, Moreno BH, Hu-Lieskovan S, Berent-Maoz B, Pang J, Chmielowski B, Cherry G, Seja E, Lomeli S, Kong X, Kelley MC, Sosman JA, Johnson DB, Ribas A, Lo RS. Genomic and Transcriptomic Features of Response to Anti-PD-1 Therapy in Metastatic Melanoma. Cell. 2017 Jan 26;168(3):542. doi: 10.1016/j.cell.2017.01.010. No abstract available. PMID 28129544
- [Background] Rayner E, van Gool IC, Palles C, Kearsey SE, Bosse T, Tomlinson I, Church DN. A panoply of errors: polymerase proofreading domain mutations in cancer. Nat Rev Cancer. 2016 Feb;16(2):71-81. doi: 10.1038/nrc.2015.12. PMID 26822575
- [Background] Church DN, Stelloo E, Nout RA, Valtcheva N, Depreeuw J, ter Haar N, Noske A, Amant F, Tomlinson IP, Wild PJ, Lambrechts D, Jurgenliemk-Schulz IM, Jobsen JJ, Smit VT, Creutzberg CL, Bosse T. Prognostic significance of POLE proofreading mutations in endometrial cancer. J Natl Cancer Inst. 2014 Dec 12;107(1):402. doi: 10.1093/jnci/dju402. Print 2015 Jan. PMID 25505230
- [Background] Johanns TM, Miller CA, Dorward IG, Tsien C, Chang E, Perry A, Uppaluri R, Ferguson C, Schmidt RE, Dahiya S, Ansstas G, Mardis ER, Dunn GP. Immunogenomics of Hypermutated Glioblastoma: A Patient with Germline POLE Deficiency Treated with Checkpoint Blockade Immunotherapy. Cancer Discov. 2016 Nov;6(11):1230-1236. doi: 10.1158/2159-8290.CD-16-0575. Epub 2016 Sep 28. PMID 27683556
- [Background] Morse CB, Elvin JA, Gay LM, Liao JB. Elevated tumor mutational burden and prolonged clinical response to anti-PD-L1 antibody in platinum-resistant recurrent ovarian cancer. Gynecol Oncol Rep. 2017 Jun 27;21:78-80. doi: 10.1016/j.gore.2017.06.013. eCollection 2017 Aug. PMID 28736741
- [Derived] Kim JW, Lee HJ, Lee JY, Park SR, Kim YJ, Hwang IG, Kyun Bae W, Byun JH, Kim JS, Kang EJ, Lee J, Shin SJ, Chang WJ, Kim EO, Sa JK, Park KH. Phase II study of nivolumab in patients with genetic alterations in DNA damage repair and response who progressed after standard treatment for metastatic solid cancers (KM-06). J Immunother Cancer. 2024 Mar 13;12(3):e008638. doi: 10.1136/jitc-2023-008638. PMID 38485184